CLINICAL TRIAL: NCT05871463
Title: Clinical Trial Phase IIa, on Amelioration of Decompensated Liver Cirrhosis With Mesenchymal Stem Cells-derived Exosomes
Brief Title: Effect of Mesenchymal Stem Cells-derived Exosomes in Decompensated Liver Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Institute for Gastroenterology and Liver Diseases (RIGLD) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1208
Record Dates: First submitted 2023-04-07; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Decompensated Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exosome (Experimental): Standard medication + MSC-derived exosomes at a final dose of 40mg in three weeks
  Interventions: Biological: MSC-derived exosomes

INTERVENTIONS:
Biological: MSC-derived exosomes — Patients will receive standard medication plus MSC-derived exosomes at a final dose of 40mg in three weeks. Standard medication includes: a) treatment of the underlying cause of cirrhosis such as drug treatment of hepatitis B and C. b) symptomatic treatment of port complications such as ascites, prevention of variceal bleeding, treatment and prevention of hepatic encephalopathy.

SUMMARY:
Decompensated liver cirrhosis (LC), a life-threatening complication of chronic liver disease, is one of the major indications for liver transplantation. Recently, mesenchymal stem cell (MSC) transfusion has been shown to lead to the regression of liver fibrosis in mice and humans. However, little is known about MSC-exosome therapy. We will evaluate the therapeutic potential of mesenchymal stem Cell-Exosomes as an alternative to cell therapy in Cirrhotic patients. This study examined the safety and efficacy of umbilical cord-derived MSC-exosomes in patients with decompensated LC.

DETAILED DESCRIPTION:
Liver fibrosis is the major cause of morbidity and mortality in patients with liver disorders. Liver fibrosis can be reverted with the removal of the underlying etiology. However, if chronic inflammation and injury persist, liver fibrosis is likely to progress to liver cirrhosis (LC). LC is generally characterized by the formation and accumulation of an extracellular matrix, which lead to the progressive distortion of the hepatic architecture. LC usually progresses irreversibly into a decompensated stage, which is characterized by a series of clinical manifestations, including ascites, variceal hemorrhage, and hepatic encephalopathy, while ascites is the most common clinical symptom in such patients. Although ascites might be treated with diuretics, periodic paracentesis, or a transjugular intrahepatic portosystemic shunt, liver transplantation is the only option that can improve the survival of these patients. However, the severe shortage of donor livers, high costs, and potential serious complications have restricted the availability of liver transplantation worldwide. Therefore, alternative strategies are under intense investigation. Mesenchymal stem cells (MSC) have self-renewal abilities and multidirectional differentiation potentials. They also interact with various types of immune cells, leading to immunomodulation. MSCs have been used therapeutically in clinical trials for graft-versus-host disease and appear to be effective in immune-mediated tissue injury, transplantation, and autoimmunity. In particular, MSCs have also been used to treat liver diseases in animal models and patients. Studies from animal models have shown that bone marrow-derived MSC (BM-MSC) infusion ameliorates liver fibrosis and reverses fulminant hepatic failure. In clinical trials, autologous MSC infusion has been demonstrated to be safe, feasible and can improve the liver function of some LC patients. In addition, BM-MSC from patients with chronic HBV infection suffer from proliferative deficiency and might not be the best choice. In contrast, human umbilical cord-derived MSC (UC-MSC) are free from these limitations related to autologous BM-MSC. In addition, UC-MSC can be obtained from the discarded UC, and therefore, can be produced on a large scale. It has been reported that human UC-MSC infusion can improve liver fibrosis in rats. It has been shown that UC-MSC have potential to be used in clinical scenarios for the treatment of human liver diseases. In the present study, the investigators examine the safety and efficacy of UC-MSC derived exosomes in decompensated LC patients. 15 enrolled patients will receive standard medication plus MSC-derived exosomes at a final dose of 40mg in three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to voluntarily sign an informed consent form (ICF) authorization.
* Males or females between 18-75 years old with a clinically confirmed diagnosis of Liver cirrhosis with any etiology, except viral cirrhosis.
* Child score class B or C.

Exclusion Criteria:

* Known cardiovascular disease.
* a) History of hepatocellular carcinoma (HCC). b) History of malignancy within the past 5 years or ongoing malignancy other than basal cell carcinoma, or resected noninvasive cutaneous squamous carcinoma at the time of Screening visit. c) Active, serious infections that require parenteral antibiotic or antifungal therapy within 30 days prior to Screening visit.
* Females who are pregnant or breastfeeding.
* Current or anticipated treatment with radiation therapy, cytotoxic chemotherapeutic agents and immunomodulating agents (such as systemic corticosteroids, interleukins, interferons).
* Use of any experimental medications within the last 6 months of Screening Visit.
* Any other clinically significant disorders or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing and protocol requirements.
* Weight loss of >5% within 6 months prior to Screening, based on subject's reporting.
* Currently or participated in a weight loss program within the last 6 months.
* Any history of bariatric surgery.
* Diabetes mellitus Type I.
* Daily alcohol intake >20 ml (2 units)/day for women and 30 ml (3 units)/day for men (on average), as per Alcohol Use Disorders Identification Test (AUDIT) questionnaire at Screening and plan to consume the same alcohol amount referenced above during the trial.
* Use of any immunosuppressive medication, anti-inflammatory monoclonal antibody treatment, or chronic systemic corticosteroids >10 mg prednisone-equivalent concurrently or within 1 year prior to Screening.
* Uncontrolled or clinically unstable thyroid disease, in the judgment of the Principal Investigator.
* Uncontrolled arterial hypertension.
* Any severe, acute, or chronic medical or psychiatric condition that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-05-26 (Estimated); Primary Completion 2023-08-11 (Estimated); Study Completion 2023-12-11 (Estimated)

PRIMARY OUTCOMES:
Liver function by MELD score | Baseline
  Calculation of MELD score based on patient's laboratory values for serum creatinine, bilirubin, international normalized ratio for prothrombin time, and sodium.
Liver function by MELD score | after 2 months of the trial
  Calculation of MELD score based on patient's laboratory values for serum creatinine, bilirubin, international normalized ratio for prothrombin time, and sodium.
Liver function by MELD score | after 4 months of the trial
  Calculation of MELD score based on patient's laboratory values for serum creatinine, bilirubin, international normalized ratio for prothrombin time, and sodium.
Liver function by CHILD score | Baseline
  Calculation of CHILD score based on patient's laboratory values for serum bilirubin, albumin, international normalized ratio for prothrombin time, ascites, and encephalopathy.
Liver function by CHILD score | after 2 months of the trial
  Calculation of CHILD score based on patient's laboratory values for serum bilirubin, albumin, international normalized ratio for prothrombin time, ascites, and encephalopathy.
Liver function by CHILD score | after 4 months of the trial
  Calculation of CHILD score based on patient's laboratory values for serum bilirubin, albumin, international normalized ratio for prothrombin time, ascites, and encephalopathy.

SECONDARY OUTCOMES:
Change in liver enzyme AST | Baseline, after 2 and 4 months of the trial
  Blood test
Change in liver enzyme ALT | Baseline, after 2 and 4 months of the trial
  Blood test
international normalized ratio (INR) for prothrombin time | Baseline, after 2 and 4 months of the trial
  Blood test
Bilirubin | Baseline, after 2 and 4 months of the trial
  Blood test

CONTACTS AND LOCATIONS:
Overall Officials: Behzad Hatami, MD, Principal Investigator — Research Institute for Gastroenterology and Liver Diseases, Shahid Beheshti Medical University, Tehran, Iran
Locations (1):
- Research Institute of Gastroenterology & Liver Diseases, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make this available.